CLINICAL TRIAL: NCT02312713
Title: Physical Therapy Versus Internet-Based Exercise Training for Patients With Knee Osteoarthritis
Acronym: PATH-IN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-1331
Record Dates: First submitted 2014-10-20; First posted 2014-12-09 (Estimated); Results first posted 2017-10-27 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-06

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard Physical Therapy (Active Comparator): Participants assigned to the PT arm will receive 3-8 individual visits with a physical therapist. The content of these visits will be "semi-standardized," meaning that they will include some common core components (e.g., evaluation, prescription of home exercise program), but the therapists will have flexibility in terms of how many visits are appropriate and the details of the visit content.
  Interventions: Behavioral: Physical Therapy
- Internet Based Exercise Training (Experimental): Participants assigned to the internet-based exercise training arm will be given access to a program that aims to tailor exercises based on individuals' functional levels. The program assigns specific exercises, progresses these exercises as appropriate over time, and shows individual video clips to demonstrate appropriate performance of exercises.
  Interventions: Behavioral: Internet Based Exercise Training
- Wait list control (No Intervention): no intervention

INTERVENTIONS:
Behavioral: Internet Based Exercise Training — Participants assigned to the PT arm will receive 3-8 individual visits with a physical therapist. The content of these visits will be "semi-standardized," meaning that they will include some common core components (e.g., evaluation, prescription of home exercise program), but the therapists will have flexibility in terms of how many visits are appropriate and the details of the visit content.
  Arms: Internet Based Exercise Training
Behavioral: Physical Therapy — Participants assigned to the internet-based exercise training arm will be given access to a program that aims to tailor exercises based on individuals' functional levels. The program assigns specific exercises, progresses these exercises as appropriate over time, and shows individual video clips to demonstrate appropriate performance of exercises.
  Arms: Standard Physical Therapy

SUMMARY:
The purpose of this study is to examine the effectiveness of standard physical therapy and an internet-based exercise program for people with knee osteoarthritis (OA). Both of these programs will be compared to a "waiting list" control group. The investigators hypothesize that both treatments will result in greater improvement than the control condition and that the treatments will be similarly effective. The investigators also expect that some patients may do better with one treatment type or another and will explore this.

ELIGIBILITY:
Inclusion Criteria:

* Knee Osteoarthritis

Exclusion Criteria:

* no internet access
* rheumatoid arthritis, lupus, or any other rheumatic condition
* severe fibromyalgia
* gout in your knees
* on a waiting list for joint replacement surgery, or are you planning to have joint replacement surgery during the next year
* total knee replacement surgery, other knee surgery, a torn meniscus in your knee, or a torn ACL in your knee during the past 6 months
* hospitalized for a stroke, heart attack, heart failure, or had surgery for blocked arteries in the past 3 months
* currently undergoing physical therapy for knee OA
* meeting current recommendations for physical activity levels
* participating in another interventional study related to knee osteoarthritis or a study that involves physical activity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2014-11; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelli D Allen, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Thurston Arthritis Research Center, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Kim S, Kosorok MR, Arbeeva L, Schwartz TA, Callahan LF, Golightly YM, Nelson AE, Allen KD. Precision Medicine-Based Machine Learning Analyses to Explore Optimal Exercise Therapies for Individuals With Knee Osteoarthritis: Random Forest-Informed Tree-Based Learning. J Rheumatol. 2023 Oct;50(10):1341-1345. doi: 10.3899/jrheum.2022-1039. Epub 2023 Aug 1. PMID 37527856
- [Derived] Coffman CJ, Arbeeva L, Schwartz TA, Callahan LF, Golightly YM, Goode AP, Huffman KM, Allen KD. Application of Heterogeneity of Treatment-Effects Methods: Exploratory Analyses of a Trial of Exercise-Based Interventions for Knee Osteoarthritis. Arthritis Care Res (Hoboken). 2022 Aug;74(8):1359-1368. doi: 10.1002/acr.24564. Epub 2022 May 2. PMID 33463020
- [Derived] Flowers PPE, Schwartz TA, Arbeeva L, Golightly YM, Pathak A, Cooke J, Gupta JJ, Callahan LF, Goode AP, Corsi M, Huffman KM, Allen KD. Racial Differences in Performance-Based Function and Potential Explanatory Factors Among Individuals With Knee Osteoarthritis. Arthritis Care Res (Hoboken). 2020 Sep;72(9):1196-1204. doi: 10.1002/acr.24018. PMID 31254451
- [Derived] Pignato M, Arbeeva L, Schwartz TA, Callahan LF, Cooke J, Golightly YM, Goode AP, Heiderscheit BC, Hill C, Huffman KM, Severson HH, Allen KD. Level of participation in physical therapy or an internet-based exercise training program: associations with outcomes for patients with knee osteoarthritis. BMC Musculoskelet Disord. 2018 Jul 19;19(1):238. doi: 10.1186/s12891-018-2139-y. PMID 30025540
- [Derived] Allen KD, Arbeeva L, Callahan LF, Golightly YM, Goode AP, Heiderscheit BC, Huffman KM, Severson HH, Schwartz TA. Physical therapy vs internet-based exercise training for patients with knee osteoarthritis: results of a randomized controlled trial. Osteoarthritis Cartilage. 2018 Mar;26(3):383-396. doi: 10.1016/j.joca.2017.12.008. Epub 2018 Jan 5. PMID 29307722
- [Derived] Gunn AH, Schwartz TA, Arbeeva LS, Callahan LF, Golightly Y, Goode A, Hill CH, Huffman K, Iversen MD, Pathak A, Taylor SS, Allen KD. Fear of Movement and Associated Factors Among Adults With Symptomatic Knee Osteoarthritis. Arthritis Care Res (Hoboken). 2017 Dec;69(12):1826-1833. doi: 10.1002/acr.23226. Epub 2017 Nov 6. PMID 28371481
- [Derived] Williams QI, Gunn AH, Beaulieu JE, Benas BC, Buley B, Callahan LF, Cantrell J, Genova AP, Golightly YM, Goode AP, Gridley CI, Gross MT, Heiderscheit BC, Hill CH, Huffman KM, Kline A, Schwartz TA, Allen KD. Physical therapy vs. internet-based exercise training (PATH-IN) for patients with knee osteoarthritis: study protocol of a randomized controlled trial. BMC Musculoskelet Disord. 2015 Sep 28;16:264. doi: 10.1186/s12891-015-0725-9. PMID 26416025

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Physical Therapy | Internet Based Exercise Training | Wait List Control
Started | 140 | 142 | 68
Completed | 129 | 112 | 63
Not Completed | 11 | 30 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Physical Therapy | Internet Based Exercise Training | Wait List Control | Total
Number analyzed (Participants) | 140 | 142 | 68 | 350
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (10.3) | 65.3 (11.5) | 64.3 (12.2) | 65.3 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 44 | 15 | 99
  Male | 100 | 98 | 53 | 251
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 1 | 9
  Not Hispanic or Latino | 134 | 138 | 67 | 339
  Unknown or Not Reported | 2 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 3
  Asian | 1 | 8 | 2 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 2
  Black or African American | 24 | 33 | 13 | 70
  White | 109 | 94 | 49 | 252
  More than one race | 1 | 2 | 1 | 4
  Unknown or Not Reported | 4 | 3 | 1 | 8
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 31.9 (8.6) | 31.5 (7.8) | 30.1 (7.3) | 31.4 (8.0)
Married or Living with Partner [Count of Participants; unit: Participants] | 80 | 93 | 42 | 215
Bachelors Degree or More Education [Count of Participants; unit: Participants] | 86 | 80 | 42 | 208
Employed [Count of Participants; unit: Participants] | 59 | 51 | 31 | 141
Low Income Financial Status [Count of Participants; unit: Participants] — "Low income" defined as self report of "just meeting basic expenses" or "don't even have enough to meet basic expenses" vs. responses of "live comfortably or "meet your basic expenses with a little left over for extras" in response to a question asking participants to "describe your household's financial situation."
  Participants | 20 | 29 | 13 | 62
Fair or Poor Self-Reported Health [Count of Participants; unit: Participants] — Participants were asked, "How would you rate your current health?" Options were: excellent, very good, good, fair and poor.
  For this metric we grouped those reporting fair or poor.
  Participants | 14 | 22 | 12 | 48
Number of Joints with Arthritis Symptoms [Mean (Standard Deviation); unit: joints] | 5.5 (3.0) | 5.2 (3.1) | 5.5 (3.9) | 5.4 (3.2)
Self-reported Years with Arthritis Symptoms [Mean (Standard Deviation); unit: years] | 14.1 (11.6) | 11.6 (11.0) | 14.2 (13.0) | 13.1 (11.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Month 4 and Change From Baseline to 12 Month in Western Ontario and McMasters Universities Osteoarthritis (WOMAC) Index Score
Description: Change over time in the primary outcome measure for this study, the WOMAC is a measure of lower extremity pain (5 items), stiffness (2 items), and function (17 items). The scale ranges from 0-96 with higher scores indicating worse symptoms and function.
Time Frame: baseline, 4 months, and 12 months
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Physical Therapy | Internet Based Exercise Training | Wait List Control
Number analyzed (Participants) | 140 | 142 | 68
units on a scale
  Baseline to 4 Month Change | -6.73 [-8.86 to -4.60] | -6.06 [-8.29 to -3.84] | -3.37 [-6.33 to -0.41]
  Baseline to 12 Month Change | -4.42 [-6.66 to -2.17] | -5.46 [-7.82 to -3.09] | -2.83 [-5.93 to 0.27]
Statistical Analysis 1: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 4 months; Test type: Superiority; p = 0.06, Mixed Models Analysis; Mean Difference (Final Values) = -3.36, 95% CI 2-sided [-6.84 to 0.12]
Statistical Analysis 2: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 12 months; Test type: Superiority; p = 0.39, Mixed Models Analysis; Mean Difference (Final Values) = -1.59, 95% CI 2-sided [-5.26 to 2.08]
Statistical Analysis 3: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 4 months; Test type: Superiority; p = 0.14, Mixed Models Analysis; Mean Difference (Final Values) = -2.70, 95% CI 2-sided [-6.24 to 0.85]
Statistical Analysis 4: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 12 months; Test type: Superiority; p = 0.17, Mixed Models Analysis; Mean Difference (Final Values) = -2.63, 95% CI 2-sided [-6.37 to 1.11]
Statistical Analysis 5: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet Based Exercise Training at 4 months; Test type: Non-Inferiority — The IBET intervention will be non-inferior to the standard PT intervention, indicated by a mean WOMAC score less than 5 points higher than standard PT; p = 0.65, Mixed Models Analysis; Mean Difference (Final Values) = 0.67, 95% CI 2-sided [-2.23 to 3.56]
Statistical Analysis 6: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet-Based Exercise Training at 12 months; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 5]; p = 0.51, Mixed Models Analysis; Mean Difference (Final Values) = -1.04, 95% CI 2-sided [-4.13 to 2.05]

2. Secondary Outcome: Change From Baseline to Month 4 and Change From Baseline to 12 Month in the Satisfaction With Physical Function Scale
Description: This is a validated, 5-item questionnaire that assesses patients' satisfaction with their ability to complete basic functional tasks that are often affected by lower extremity OA, including stair-climbing, walking, doing housework (light and heavy, and lifting and carrying). All 5 items are rated on a 7 point scale ranging from Very Dissatisfied (-3) Very Satisfied (+3). The total scale ranges from -15 to +15,with higher scores indicating greater satisfaction with function.
Time Frame: baseline, 4 months, and 12 months
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Physical Therapy | Internet Based Exercise Training | Wait List Control
Number analyzed (Participants) | 140 | 142 | 68
units on a scale
  Baseline to 4 Month Change | 0.84 [0.6 to 1.09] | 0.35 [0.09 to 0.61] | 0.28 [-0.07 to 0.63]
  Baseline to 12 Month Change | 0.39 [0.14 to 0.64] | 0.43 [0.16 to 0.70] | 0.16 [-0.19 to 0.51]
Statistical Analysis 1: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 4 months; Test type: Superiority; p = 0.01, Mixed Models Analysis; Median Difference (Final Values) = 0.56, 95% CI 2-sided [0.15 to 0.98]
Statistical Analysis 2: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 12 months; Test type: Superiority; p = 0.28, Mixed Models Analysis; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-0.19 to 0.65]
Statistical Analysis 3: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 4 months; Test type: Superiority; p = 0.75, Mixed Models Analysis; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.35 to 0.49]
Statistical Analysis 4: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 12 months; Test type: Superiority; p = 0.22, Mixed Models Analysis; Mean Difference (Final Values) = 0.27, 95% CI 2-sided [-0.16 to 0.7]
Statistical Analysis 5: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet Based Exercise Training at 4 months; Test type: Non-Inferiority — Since there were not sufficient data in prior literature to specific an a priori non-inferiority margin, for this and other secondary outcomes we based conclusions and discussions on magnitude of differences between the group, descriptively. This strategy was specified in the protocol; p = 0.00, Mixed Models Analysis; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.84 to -0.16]
Statistical Analysis 6: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet-Based Exercise Training at 12 months; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = 0.83, Mixed Models Analysis; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.31 to 0.39]

3. Secondary Outcome: Change From Baseline to Month 4 and Change From Baseline to 12 Month in Objective Physical Function - 2 Minute Step Test
Description: One of 4 tests that objectively assessed physical function. These 4 tests included: unilateral stand time; time to rise from a chair and return to the seated position for 30 seconds; timed up and go- rise from a seated position, walk a short distance and return to seated position; and a 2 minute step test. For this outcome measure, the 2 minute step test, the minimum is 0 steps and there is no maximum scale score (participants complete as many steps as they can in 2 minutes); greater steps indicate better function.
Time Frame: baseline, 4 months, and 12 months
Measure: Least Squares Mean (95% Confidence Interval); unit: number of steps taken in 2 minutes
Arm/Group | Standard Physical Therapy | Internet Based Exercise Training | Wait List Control
Number analyzed (Participants) | 140 | 142 | 68
number of steps taken in 2 minutes
  Baseline to 4 Month Change | -0.68 [-5.07 to 3.71] | -3.54 [-8.20 to 1.11] | -8.43 [-14.61 to -2.24]
  Baseline to 12 Month Change | 1.11 [-3.45 to 5.67] | 1.12 [-3.76 to 6] | 0.00 [-6.49 to 6.48]
Statistical Analysis 1: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 4 months for the 2 Minute Step Test; Test type: Superiority; p = 0.04, Mixed Models Analysis; Mean Difference (Final Values) = 7.75, 95% CI 2-sided [0.43 to 15.07]
Statistical Analysis 2: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 12 months for the 2 Minute Step Test; Test type: Superiority; p = 0.78, Mixed Models Analysis; Mean Difference (Final Values) = 1.12, 95% CI 2-sided [-6.59 to 8.82]
Statistical Analysis 3: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 4 months for the 2 Minute Step Test; Test type: Superiority; p = 0.20, Mixed Models Analysis; Mean Difference (Final Values) = 4.88, 95% CI 2-sided [-2.56 to 12.33]
Statistical Analysis 4: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 12 months for the 2 Minute Step Test; Test type: Superiority; p = .78, Mixed Models Analysis; Mean Difference (Final Values) = 1.13, 95% CI 2-sided [-6.74 to 8.99]
Statistical Analysis 5: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet Based Exercise Training at 4 months for the 2 Minute Step Test; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = 0.35, Mixed Models Analysis; Mean Difference (Final Values) = -2.86, 95% CI 2-sided [-8.94 to 3.21]
Statistical Analysis 6: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet Based Exercise Training at 12 months for the 2 Minute Step Test; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = 1.00, Mixed Models Analysis; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-6.40 to 6.42]

4. Secondary Outcome: Change From Baseline to Month 4 and Change From Baseline to 12 Month in Objective Physical Function- Unilateral Stand Time
Description: One of 4 tests that objectively assessed physical function. These 4 tests included: unilateral stand time; time to rise from a chair and return to the seated position for 30 seconds; timed up and go- rise from a seated position, walk a short distance and return to seated position; and a 2 minute step test. For this outcome measure, the unilateral stand test, scores scan range from 0-10 seconds, with higher time indicating better balance.
Time Frame: baseline, 4 months, and 12 months
Measure: Least Squares Mean (95% Confidence Interval); unit: seconds
Arm/Group | Standard Physical Therapy | Internet Based Exercise Training | Wait List Control
Number analyzed (Participants) | 140 | 142 | 68
seconds
  Baseline to 4 Month Change | -0.59 [-1.15 to -0.03] | 0.02 [-0.57 to 0.61] | 0.04 [-0.75 to 0.82]
  Baseline to 12 Month Change | -0.05 [-0.6 to 0.50] | -0.05 [-0.64 to 0.53] | -0.09 [-0.88 to 0.69]
Statistical Analysis 1: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 4 months for Unilateral Stand Time; Test type: Superiority; p = 0.19, Mixed Models Analysis; Mean Difference (Final Values) = -0.63, 95% CI 2-sided [-1.56 to 0.30]
Statistical Analysis 2: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 12 months for Unilateral Stand Time; Test type: Superiority; p = 0.93, Mixed Models Analysis; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.89 to 0.98]
Statistical Analysis 3: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 4 months for Unilateral Stand Time; Test type: Superiority; p = 0.97, Mixed Models Analysis; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.97 to 0.93]
Statistical Analysis 4: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 12 months for Unilateral Stand Time; Test type: Superiority; p = 0.93, Mixed Models Analysis; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.91 to 1]
Statistical Analysis 5: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet Based Exercise Training at 4 months for Unilateral Stand Time; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = 0.12, Mixed Models Analysis; Mean Difference (Final Values) = 0.61, 95% CI 2-sided [-0.16 to 1.38]
Statistical Analysis 6: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet Based Exercise Training at 12 months for Unilateral Stand Time; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = 1.00, Mixed Models Analysis; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.78 to 0.77]

5. Secondary Outcome: Change From Baseline to Month 4 and Change From Baseline to 12 Month in Objective Physical Function - 30 Second Chair Stand
Description: One of 4 tests that objectively assessed physical function. These 4 tests included: unilateral stand time; time to rise from a chair and return to the seated position for 30 seconds; timed up and go- rise from a seated position, walk a short distance and return to seated position; and a 2 minute step test. For this outcome measure, the 30 second chair stand test, the minimum is 0 stands and there is no maximum scale score (participants complete as many stands as they can in 30 seconds; greater numbers of stands indicate better function.
Time Frame: baseline, 4 months, and 12 months
Measure: Least Squares Mean (95% Confidence Interval); unit: number of stands from a chair in 30 sec
Arm/Group | Standard Physical Therapy | Internet Based Exercise Training | Wait List Control
Number analyzed (Participants) | 140 | 142 | 68
number of stands from a chair in 30 sec
  Baseline to 4 Month Change | -0.13 [-0.87 to 0.61] | 0.50 [-0.29 to 1.28] | 0.18 [-0.87 to 1.23]
  Baseline to 12 Month Change | 0.16 [-0.49 to 0.82] | 0.90 [0.20 to 1.60] | 0.66 [-0.27 to 1.58]
Statistical Analysis 1: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 4 months for 30 Second Chair Stand; Test type: Superiority; p = 0.63, Mixed Models Analysis; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-1.55 to .94]
Statistical Analysis 2: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 12 months for 30 Second Chair Stand; Test type: Superiority; p = 0.37, Mixed Models Analysis; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-1.58 to 0.6]
Statistical Analysis 3: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 4 months for 30 Second Chair Stand; Test type: Superiority; p = 0.62, Mixed Models Analysis; Mean Difference (Final Values) = 0.32, 95% CI 2-sided [-0.95 to 1.59]
Statistical Analysis 4: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 12 months for 30 Second Chair Stand; Test type: Superiority; p = 0.67, Mixed Models Analysis; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-0.87 to 1.35]
Statistical Analysis 5: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet Based Exercise Training at 4 months for 30 Second Chair Stand; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = 0.23, Mixed Models Analysis; Mean Difference (Final Values) = 0.63, 95% CI 2-sided [-0.40 to 1.66]
Statistical Analysis 6: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet Based Exercise Training at 12 months for 30 Second Chair Stand; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = 0.11, Mixed Models Analysis; Mean Difference (Final Values) = 0.74, 95% CI 2-sided [-0.17 to 1.64]

6. Secondary Outcome: Change From Baseline to Month 4 and Change From Baseline to 12 Month in Objective Physical Function- Timed Up and Go
Description: One of 4 tests that objectively assessed physical function. These 4 tests included: unilateral stand time; time to rise from a chair and return to the seated position for 30 seconds; timed up and go- rise from a seated position, walk a short distance and return to seated position; and a 2 minute step test. For this outcome measure, the timed up and go, there are no minimum or maximum scores (participants complete the task as quickly as they are able); shorter (lower) times indicate better function.
Time Frame: baseline, 4 months, and 12 months
Measure: Least Squares Mean (95% Confidence Interval); unit: seconds
Arm/Group | Standard Physical Therapy | Internet Based Exercise Training | Wait List Control
Number analyzed (Participants) | 140 | 142 | 68
seconds
  Baseline to 4 Month Change | -0.62 [-1.34 to 0.09] | -0.87 [-1.63 to -0.11] | -0.23 [-1.24 to 0.78]
  Baseline to 12 Month Change | -0.77 [-1.57 to 0.04] | -1.49 [-2.35 to -0.63] | -0.26 [-1.4 to 0.87]
Statistical Analysis 1: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 4 months for Timed Up and Go; Test type: Superiority; p = 0.52, Mixed Models Analysis; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-1.58 to 0.8]
Statistical Analysis 2: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 12 months for Timed Up and Go; Test type: Superiority; p = 0.46, Mixed Models Analysis; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.86 to 0.85]
Statistical Analysis 3: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 4 months for Timed Up and Go; Test type: Superiority; p = 0.3, Mixed Models Analysis; Mean Difference (Final Values) = -0.64, 95% CI 2-sided [-1.85 to 0.58]
Statistical Analysis 4: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 12 months for Timed Up and Go; Test type: Superiority; p = 0.08, Mixed Models Analysis; Mean Difference (Final Values) = -1.22, 95% CI 2-sided [-2.61 to 0.16]
Statistical Analysis 5: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet Based Exercise Training at 4 months for Timed Up and Go; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = 0.63, Mixed Models Analysis; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-1.23 to 0.74]
Statistical Analysis 6: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet Based Exercise Training at 12 months for Timed Up and Go; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = 0.21, Mixed Models Analysis; Mean Difference (Final Values) = -0.72, 95% CI 2-sided [-1.85 to 0.41]

7. Secondary Outcome: Change From Baseline to Month 4 and Change From Baseline to 12 Month in the Patient Health Questionnaire-8
Description: Depressive symptoms and severity will be assessed using the PHQ-8, a reliable and valid measure of depression71. The PHQ-8 is an eight-item survey derived from the Primary Care Evaluation of Mental Disorders (PRIME-MD) diagnostic tool, and consists of items corresponding to the depression criteria listed in the Diagnostic and Statistics Manual Fourth Edition (DSM-IV). Each of the eight questions is scored as 0 (not at all) to 3 (nearly every day), so that total scores range from 0 to 24, with higher scores indicating more depressive symptoms.
Time Frame: baseline, 4 months, and 12 months
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Physical Therapy | Internet Based Exercise Training | Wait List Control
Number analyzed (Participants) | 140 | 142 | 68
units on a scale
  Baseline to 4 Month Change | -0.46 [-0.94 to 0.02] | -0.22 [-0.73 to 0.29] | 0.33 [-0.36 to 1.01]
  Baseline to 12 Month Change | 0.1 [-0.45 to 0.65] | 0.1 [-0.49 to 0.69] | 0.99 [0.22 to 1.77]
Statistical Analysis 1: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 4 months; Test type: Superiority; p = 0.05, Mixed Models Analysis; Mean Difference (Final Values) = -0.79, 95% CI 2-sided [-1.59 to 0.02]
Statistical Analysis 2: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 12 months; Test type: Superiority; p = 0.05, Mixed Models Analysis; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.82 to 0.02]
Statistical Analysis 3: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 4 months; Test type: Superiority; p = 0.19, Mixed Models Analysis; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-1.37 to 0.27]
Statistical Analysis 4: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 12 months; Test type: Superiority; p = 0.06, Mixed Models Analysis; Mean Difference (Final Values) = -0.89, 95% CI 2-sided [-1.83 to 0.05]
Statistical Analysis 5: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet Based Exercise Training at 4 months; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = 0.49, Mixed Models Analysis; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-0.43 to 0.89]
Statistical Analysis 6: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet-Based Exercise Training at 12 months; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = 0.99, Mixed Models Analysis; Mean Difference (Final Values) = 0, 95% CI 2-sided [-0.77 to 0.78]

8. Secondary Outcome: Change From Baseline to Month 4 and Change From Baseline to Month 12 in The Knee Injury and Osteoarthritis Outcome Score (KOOS)
Description: The KOOS is a patient-reported outcome measurement instrument, developed to assess the patient's opinion about their knee and associated problems. Five KOOS subscale scores were administered: Pain (9 items), Function in daily living (17 items), Function in Sport and Recreation (5 items), and knee-related Quality of Life (4 items). All items are scored on 5-point Likert scales. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale
Time Frame: baseline, 4 months, and 12 months
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Physical Therapy | Internet Based Exercise Training | Wait List Control
Number analyzed (Participants) | 140 | 142 | 68
units on a scale
  Baseline to 4 Month Change - KOOS Pain | 6.2 [3.75 to 8.65] | 7.77 [5.17 to 10.38] | 3.84 [0.38 to 7.29]
  Baseline to 12 Month Change - KOOS Pain | 3.67 [1.05 to 6.29] | 6.18 [3.38 to 8.98] | 2.82 [-0.86 to 6.5]
  Baseline to 4 Month Change - KOOS ADL | 6.8 [4.53 to 9.06] | 5.47 [3.08 to 7.87] | 3.37 [0.16 to 6.57]
  Baseline to 12 Month Change - KOOS ADL | 4.65 [2.3 to 7.01] | 4.99 [2.48 to 7.49] | 2.2 [-1.1 to 5.5]
  Baseline to 4 Month Change - KOOS Sport/Rec | 5.6 [2.44 to 8.77] | 5.4 [2.03 to 8.77] | 1.69 [-2.82 to 6.2]
  Baseline to 12 Month Change - KOOS Sport/Rec | 5.44 [2.07 to 8.8] | 5.98 [2.33 to 9.64] | -0.03 [-4.76 to 4.7]
  Baseline to 4 Month Change - KOOS QOL | 5.56 [2.93 to 8.19] | 5.9 [3.11 to 8.69] | 2.27 [-1.45 to 5.99]
  Baseline to 12 Month Change - KOOS QOL | 4.21 [1.64 to 6.78] | 6.8 [4.06 to 9.54] | -0.93 [-4.53 to 2.66]
Statistical Analysis 1: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet Based Exercise Training at 4 months for KOOS Pain; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = 0.36, Mixed Models Analysis; Mean Difference (Final Values) = 1.57, 95% CI 2-sided [-1.77 to 4.92]
Statistical Analysis 2: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet-Based Exercise Training at 12 months for KOOS Pain; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = 0.17, Mixed Models Analysis; Mean Difference (Final Values) = 2.51, 95% CI 2-sided [-1.11 to 6.14]
Statistical Analysis 3: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 4 months for KOOS Pain; Test type: Superiority; p = 0.06, Mixed Models Analysis; Mean Difference (Final Values) = 3.94, 95% CI 2-sided [-0.19 to 8.06]
Statistical Analysis 4: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 12 months for KOOS Pain; Test type: Superiority; p = 0.14, Mixed Models Analysis; Mean Difference (Final Values) = 3.36, 95% CI 2-sided [-1.08 to 7.79]
Statistical Analysis 5: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Standard Physical Therapy and Wait List Control at 4 months for KOOS Pain; Test type: Superiority; p = 0.25, Mixed Models Analysis; Mean Difference (Final Values) = 2.37, 95% CI 2-sided [-1.67 to 6.4]
Statistical Analysis 6: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Standard Physical Therapy and Wait List Control at 12 months for KOOS Pain; Test type: Superiority; p = 0.70, Mixed Models Analysis; Mean Difference (Final Values) = 0.85, 95% CI 2-sided [-3.48 to 5.18]
Statistical Analysis 7: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet Based Exercise Training at 4 months for KOOS ADL; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = 0.40, Mixed Models Analysis; Mean Difference (Final Values) = -1.32, 95% CI 2-sided [-4.43 to 1.79]
Statistical Analysis 8: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet Based Exercise Training at 12 months for KOOS ADL; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = 0.84, Mixed Models Analysis; Mean Difference (Final Values) = 0.33, 95% CI 2-sided [-2.93 to 3.59]
Statistical Analysis 9: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 4 month for KOOS ADL; Test type: Superiority; p = 0.28, Mixed Models Analysis; Mean Difference (Final Values) = 2.11, 95% CI 2-sided [-1.73 to 5.94]
Statistical Analysis 10: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 12 month for KOOS ADL; Test type: Superiority; p = 0.17, Mixed Models Analysis; Mean Difference (Final Values) = 2.79, 95% CI 2-sided [-1.2 to 6.77]
Statistical Analysis 11: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 4 months for KOOS ADL; Test type: Superiority; p = 0.07, Mixed Models Analysis; Mean Difference (Final Values) = 3.43, 95% CI 2-sided [-0.32 to 7.18]
Statistical Analysis 12: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 12 months for KOOS ADL; Test type: Superiority; p = 0.22, Mixed Models Analysis; Mean Difference (Final Values) = 2.45, 95% CI 2-sided [-1.44 to 6.34]
Statistical Analysis 13: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet Based Exercise Training at 4 months for KOOS Sport/Rec; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = .92, Mixed Models Analysis; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-4.47 to 4.06]
Statistical Analysis 14: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet Based Exercise Training at 12 months for KOOS Sport/Rec; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = .82, Mixed Models Analysis; Mean Difference (Final Values) = .55, 95% CI 2-sided [-4.15 to 5.24]
Statistical Analysis 15: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 4 months for KOOS Sport/Rec; Test type: Superiority; p = 0.17, Mixed Models Analysis; Mean Difference (Final Values) = 3.71, 95% CI 2-sided [-1.59 to 9]
Statistical Analysis 16: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 12 months for KOOS Sport/Rec; Test type: Superiority; p = 0.04, Mixed Models Analysis; Mean Difference (Final Values) = 6.01, 95% CI 2-sided [0.29 to 11.74]
Statistical Analysis 17: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 4 months for KOOS Sport/Rec; Test type: Superiority; p = 0.14, Mixed Models Analysis; Mean Difference (Final Values) = 3.91, 95% CI 2-sided [-1.28 to 9.1]
Statistical Analysis 18: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 12 months for KOOS Sport/Rec; Test type: Superiority; p = 0.05, Mixed Models Analysis; Mean Difference (Final Values) = 5.47, 95% CI 2-sided [-0.1 to 11.03]
Statistical Analysis 19: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet Based Exercise Training at 4 months for KOOS QOL; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = .86, Mixed Models Analysis; Mean Difference (Final Values) = .33, 95% CI 2-sided [-3.29 to 3.96]
Statistical Analysis 20: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet Based Exercise Training at 12 months for KOOS QOL; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = 0.15, Mixed Models Analysis; Mean Difference (Final Values) = 2.59, 95% CI 2-sided [-0.96 to 6.13]
Statistical Analysis 21: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 4 months for KOOS QOL; Test type: Superiority; p = 0.11, Mixed Models Analysis; Mean Difference (Final Values) = 3.63, 95% CI 2-sided [-0.85 to 8.11]
Statistical Analysis 22: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 12 months for KOOS QOL; Test type: Superiority; p = 0, Mixed Models Analysis; Mean Difference (Final Values) = 7.74, 95% CI 2-sided [3.39 to 12.08]
Statistical Analysis 23: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 4 months for KOOS QOL; Test type: Superiority; p = 0.14, Mixed Models Analysis; Mean Difference (Final Values) = 3.29, 95% CI 2-sided [-1.08 to 7.67]
Statistical Analysis 24: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 12 months for KOOS QOL; Test type: Superiority; p = 0.02, Mixed Models Analysis; Mean Difference (Final Values) = 5.15, 95% CI 2-sided [0.92 to 9.37]

9. Secondary Outcome: Change From Baseline to Month 4 and Change From Baseline to 12 Month in The PROMIS Sleep-related Impairment Instrument
Description: The PROMIS adult sleep related impairment item bank focuses on self-reported perceptions of alertness, sleepiness, and tiredness during usual waking hours, and the perceived functional impairments during wakefulness associated with sleep problems or impaired alertness. It assesses sleep-related impairment over the past seven days. This scale includes 8 items, each measured on a 5-point Likert scale. Per PROMIS scoring instructions, raw scores are converted into standardized t-scores with a mean of 50 and standard deviation of 10. T-scores can range from 30.5-77.6; higher scores indicate worse sleep impairment.
Time Frame: baseline, 4 months, and 12 months
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Physical Therapy | Internet Based Exercise Training | Wait List Control
Number analyzed (Participants) | 140 | 142 | 68
units on a scale
  Baseline to 4 Month Change | -3.13 [-4.37 to -1.89] | -0.94 [-2.26 to 0.38] | -0.54 [-2.32 to 1.23]
  Baseline to 12 Month Change | -2.16 [-3.47 to -0.86] | -0.45 [-1.84 to 0.94] | -1.1 [-2.93 to 0.72]
Statistical Analysis 1: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 4 months; Test type: Superiority; p = 0.02, Mixed Models Analysis; Mean Difference (Final Values) = -2.58, 95% CI 2-sided [-4.67 to -0.5]
Statistical Analysis 2: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 12 months; Test type: Superiority; p = 0.33, Mixed Models Analysis; Mean Difference (Final Values) = -1.06, 95% CI 2-sided [-3.22 to 1.09]
Statistical Analysis 3: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 4 months; Test type: Superiority; p = 0.72, Mixed Models Analysis; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-2.52 to 1.74]
Statistical Analysis 4: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 12 months; Test type: Superiority; p = 0.56, Mixed Models Analysis; Mean Difference (Final Values) = 0.65, 95% CI 2-sided [-1.56 to 2.86]
Statistical Analysis 5: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet Based Exercise Training at 4 months; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = 0.01, Mixed Models Analysis; Mean Difference (Final Values) = 2.19, 95% CI 2-sided [0.48 to 3.9]
Statistical Analysis 6: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet-Based Exercise Training at 12 months; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = 0.06, Mixed Models Analysis; Mean Difference (Final Values) = 1.71, 95% CI 2-sided [-0.1 to 3.52]

10. Secondary Outcome: Change From Baseline to Month 4 and Change From Baseline to 12 Month in The PROMIS Fatigue Instrument
Description: The PROMIS Fatigue instruments evaluate a range of self-reported symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles. Fatigue is divided into the experience of fatigue (frequency, duration, and intensity) and the impact of fatigue on physical, mental, and social activities. It assesses fatigue over the past seven days, This scale includes 8 items, each measured on a 5-point Likert scale. Per PROMIS scoring instructions, raw scores are converted into standardized t-scores with a mean of 50 and standard deviation of 10. T-scores can range from 33.1-77.8; higher scores indicate worse fatigue.
Time Frame: baseline, 4 months, and 12 months
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Physical Therapy | Internet Based Exercise Training | Wait List Control
Number analyzed (Participants) | 140 | 142 | 68
units on a scale
  Baseline to 4 Month Change | -0.91 [-2.21 to 0.38] | 0.57 [-0.81 to 1.94] | 1.55 [0.31 to 3.42]
  Baseline to 12 Month Change | 0.09 [-1.05 to 1.24] | 0.88 [-0.35 to 2.1] | 2.52 [0.93 to 4.12]
Statistical Analysis 1: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 4 months; Test type: Superiority; p = 0.03, Mixed Models Analysis; Mean Difference (Final Values) = -2.47, 95% CI 2-sided [-4.67 to -0.26]
Statistical Analysis 2: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 12 months; Test type: Superiority; p = 0.01, Mixed Models Analysis; Mean Difference (Final Values) = -2.43, 95% CI 2-sided [-4.31 to -0.55]
Statistical Analysis 3: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 4 months; Test type: Superiority; p = 0.39, Mixed Models Analysis; Mean Difference (Final Values) = -0.99, 95% CI 2-sided [-3.24 to 1.27]
Statistical Analysis 4: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 12 months; Test type: Superiority; p = 0.1, Mixed Models Analysis; Mean Difference (Final Values) = -1.65, 95% CI 2-sided [-3.58 to 0.29]
Statistical Analysis 5: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet Based Exercise Training at 4 months; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = 0.11, Mixed Models Analysis; Mean Difference (Final Values) = 1.48, 95% CI 2-sided [-0.33 to 3.29]
Statistical Analysis 6: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet-Based Exercise Training at 12 months; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = 0.33, Mixed Models Analysis; Mean Difference (Final Values) = 0.79, 95% CI 2-sided [-0.8 to 2.37]

11. Secondary Outcome: Change From Baseline to Month 4 and Change From Baseline to 12 Month in the The Brief Fear of Movement Scale
Description: The Brief Fear of Movement Scale is a six item scale for assessing fear of movement in OA. The scale specifically assesses activity avoidance due to pain-related fear of movement. All items are measured on a 4-point scale from "strongly agree" to "strongly disagree." The score ranges from 0-24 with higher scores indicating more fear of movement.
Time Frame: baseline, 4 months, and 12 months
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Physical Therapy | Internet Based Exercise Training | Wait List Control
Number analyzed (Participants) | 140 | 142 | 68
units on a scale
  Baseline to 4 Month Change | -0.34 [-0.84 to 0.15] | 0.01 [-0.52 to 0.53] | 0.45 [-0.26 to 1.15]
  Baseline to 12 Month Change | 0.28 [-0.19 to 0.74] | 0.06 [-0.44 to 0.56] | 0.28 [-0.37 to 0.93]
Statistical Analysis 1: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 4 months; Test type: Superiority; p = 0.06, Mixed Models Analysis; Mean Difference (Final Values) = -0.79, 95% CI 2-sided [-1.62 to 0.04]
Statistical Analysis 2: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 12 months; Test type: Superiority; p = 1.00, Mixed Models Analysis; Mean Difference (Net) = 0, 95% CI 2-sided [-0.77 to 0.77]
Statistical Analysis 3: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 4 months; Test type: Superiority; p = 0.31, Mixed Models Analysis; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-1.29 to 0.41]
Statistical Analysis 4: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 12 months; Test type: Superiority; p = 0.58, Mixed Models Analysis; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-1.01 to 0.57]
Statistical Analysis 5: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet Based Exercise Training at 4 months; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = 0.32, Mixed Models Analysis; Mean Difference (Final Values) = 0.35, 95% CI 2-sided [-0.33 to 1.03]
Statistical Analysis 6: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet-Based Exercise Training at 12 months; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = 0.51, Mixed Models Analysis; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.86 to 0.43]

12. Secondary Outcome: Change From Baseline to Month 4 and Change From Baseline to 12 Month in the Physical Activity Scale for the Elderly (PASE)
Description: The Physical Activity Scale for the Elderly (PASE) is a self-report, 12-item scale that measures level occupational, household, and leisure activity during a one-week period. This scale was particularly developed for use among older adults; although all participants in the proposed study will not be age 65 or over, patients with knee OA typically have more limited physical activity than the general population. Therefore we believe this scale will be more applicable to our participant group than scales that were developed for younger adults.
  The typical range for the total PASE score is 0-400, with higher scores indicating greater activity.
Time Frame: baseline, 4 months, and 12 months
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Physical Therapy | Internet Based Exercise Training | Wait List Control
Number analyzed (Participants) | 140 | 142 | 68
units on a scale
  Baseline to 4 Month Change | 2.25 [-9.18 to 13.68] | -11.52 [-23.79 to 0.74] | -4.7 [-21.04 to 11.64]
  Baseline to 12 Month Change | 8.28 [-2.01 to 18.56] | 8.19 [-2.99 to 19.37] | 1.17 [-13.11 to 15.45]
Statistical Analysis 1: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 4 months; Test type: Superiority; p = 0.48, Mixed Models Analysis; Mean Difference (Final Values) = 6.95, 95% CI 2-sided [-12.31 to 26.22]
Statistical Analysis 2: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 12 months; Test type: Superiority; p = 0.41, Mixed Models Analysis; Mean Difference (Final Values) = 7.11, 95% CI 2-sided [-9.69 to 23.91]
Statistical Analysis 3: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 4 months; Test type: Superiority; p = 0.50, Mixed Models Analysis; Mean Difference (Final Values) = -6.82, 95% CI 2-sided [-26.55 to 12.91]
Statistical Analysis 4: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 12 months; Test type: Superiority; p = 0.43, Mixed Models Analysis; Mean Difference (Final Values) = 7.02, 95% CI 2-sided [-10.31 to 24.35]
Statistical Analysis 5: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet Based Exercise Training at 4 months; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = 0.09, Mixed Models Analysis; Mean Difference (Final Values) = -13.77, 95% CI 2-sided [-29.73 to 2.19]
Statistical Analysis 6: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet-Based Exercise Training at 12 months; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = 0.99, Mixed Models Analysis; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-14.41 to 14.23]

13. Secondary Outcome: Change From Baseline to Month 4 and Change From Baseline to 12 Month in Additional Self-Report Physical Activity Items
Description: Number of minutes per week, on average, they are completing strengthening, stretching, and aerobic exercises. The minimum score is 0, and there is no maximum score; higher scores indicate more weekly activity.
Time Frame: baseline, 4 months, and 12 months
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes per week
Arm/Group | Standard Physical Therapy | Internet Based Exercise Training | Wait List Control
Number analyzed (Participants) | 140 | 142 | 68
minutes per week
  Baseline to 4 Month Change - Strengthening Exercis | 1.78 [0.99 to 2.57] | 1.27 [0.44 to 2.11] | 0.43 [-0.69 to 1.54]
  Baseline to 12 Month Change - Strengthening Exerc | 1.07 [0.23 to 1.91] | 1.21 [0.32 to 2.1] | -0.14 [-1.32 to 1.04]
  Baseline to 4 Month Change - Stretching | 1.45 [0.76 to 2.15] | 0.97 [0.23 to 1.72] | -0.4 [-1.39 to 0.6]
  Baseline to 12 Month Change - Stretching | 0.27 [-0.37 to 0.92] | 0.72 [0.04 to 1.41] | -1.34 [-2.24 to -0.44]
  Baseline to 4 Month Change - Aerobic Exercises | 1 [-0.02 to 2.02] | 1.79 [0.71 to 2.88] | -0.09 [-1.53 to 1.35]
  Baseline to 12 Month Change - Aerobic Exercises | 0.48 [-0.67 to 1.63] | 0.41 [-0.82 to 1.63] | -1.59 [-3.21 to 0.04]
Statistical Analysis 1: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 4 months for Strengthening Exercises; Test type: Superiority; p = 0.04, Mixed Models Analysis; Mean Difference (Final Values) = 1.36, 95% CI 2-sided [0.05 to 2.66]
Statistical Analysis 2: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 12 months for Strengthening Exercises; Test type: Superiority; p = 0.09, Mixed Models Analysis; Mean Difference (Final Values) = 1.21, 95% CI 2-sided [-0.18 to 2.6]
Statistical Analysis 3: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 4 months for Strengthening Exercises; Test type: Superiority; p = 0.22, Mixed Models Analysis; Mean Difference (Final Values) = 0.85, 95% CI 2-sided [-0.49 to 2.19]
Statistical Analysis 4: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 12 months for Strengthening Exercises; Test type: Superiority; p = 0.06, Mixed Models Analysis; Mean Difference (Final Values) = 1.35, 95% CI 2-sided [-0.08 to 2.78]
Statistical Analysis 5: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet Based Exercise Training at 4 months for Strength; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = 0.36, Mixed Models Analysis; Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-1.6 to 0.58]
Statistical Analysis 6: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet Based Exercise Training at 12 months for Strength; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = 0.81, Mixed Models Analysis; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-1.03 to 1.31]
Statistical Analysis 7: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 4 months for Stretching; Test type: Superiority; p = 0.00, Mixed Models Analysis; Mean Difference (Final Values) = 1.85, 95% CI 2-sided [0.67 to 3.03]
Statistical Analysis 8: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 12 months for Stretching; Test type: Superiority; p = 0.00, Mixed Models Analysis; Mean Difference (Final Values) = 1.62, 95% CI 2-sided [0.55 to 2.68]
Statistical Analysis 9: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 4 months for Stretching; Test type: Superiority; p = 0.03, Mixed Models Analysis; Mean Difference (Final Values) = 1.37, 95% CI 2-sided [0.16 to 2.57]
Statistical Analysis 10: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 12 months for Stretching; Test type: Superiority; p = 0.00, Mixed Models Analysis; Mean Difference (Final Values) = 2.07, 95% CI 2-sided [0.98 to 3.16]
Statistical Analysis 11: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet Based Exercise Training at 4 months for Stretching; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = 0.33, Mixed Models Analysis; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-1.46 to 0.5]
Statistical Analysis 12: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet Based Exercise Training at 12 months for Stretching; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = 0.32, Mixed Models Analysis; Mean Difference (Final Values) = 0.45, 95% CI 2-sided [-0.44 to 1.34]
Statistical Analysis 13: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 4 months for Aerobic Exercise; Test type: Superiority; p = 0.21, Mixed Models Analysis; Mean Difference (Final Values) = 1.09, 95% CI 2-sided [-0.61 to 2.8]
Statistical Analysis 14: Comparison: Standard Physical Therapy vs Wait List Control; This is the comparison between Physical Therapy and Wait List Control at 12 months for Aerobic Exercise; Test type: Superiority; p = 0.04, Mixed Models Analysis; Mean Difference (Final Values) = 2.07, 95% CI 2-sided [0.13 to 4]
Statistical Analysis 15: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 4 months for Aerobic Exercise; Test type: Superiority; p = 0.03, Mixed Models Analysis; Mean Difference (Final Values) = 1.89, 95% CI 2-sided [0.15 to 3.62]
Statistical Analysis 16: Comparison: Internet Based Exercise Training vs Wait List Control; This is the comparison between Internet Based Exercise Training and Wait List Control at 12 months for Aerobic Exercise; Test type: Superiority; p = 0.05, Mixed Models Analysis; Mean Difference (Final Values) = 1.99, 95% CI 2-sided [0.01 to 3.97]
Statistical Analysis 17: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet Based Exercise Training at 4 months for Aerobic Exercise; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = 0.27, Mixed Models Analysis; Mean Difference (Final Values) = 0.79, 95% CI 2-sided [-0.62 to 2.2]
Statistical Analysis 18: Comparison: Standard Physical Therapy vs Internet Based Exercise Training; This is the comparison between Physical Therapy and Internet Based Exercise Training at 12 months for Aerobic Exercise; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 5]; p = 0.93, Mixed Models Analysis; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-1.69 to 1.54]

ADVERSE EVENTS:
Time Frame: Data were collected for 12 months, ending at participants' final follow up time point.
Arm/Group | Standard Physical Therapy | Internet Based Exercise Training | Wait List Control
All-Cause Mortality (participants affected / at risk) | 0/140 | 2/142 | 0/68
Serious Adverse Events (participants affected / at risk) | 8/140 | 12/142 | 9/68
Other Adverse Events (participants affected / at risk) | 0/140 | 0/142 | 0/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Physical Therapy (N=140) | Internet Based Exercise Training (N=142) | Wait List Control (N=68)
Osteomyelitis of left foot (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Chronic Leukemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Embolism (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Shortness of breath, CHF exacerbation, pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Left femoral hernia resulting in small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Posterior Lumbar Decompression & Fusion Surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Heart Blockage (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Stage 1 Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Total Knee Replacement (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Heart Attack (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Cataract Surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pacemaker implant for Sick sinus syndrome (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) — with symptomatic bradycardia
Odontoid fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Asthma Exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sepsis from E.Coli UTI (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
C1 Cervical Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Laproscopy w/total hysterectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Laparoscopic cholecystectomy for cholelithiasis (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Appendicitis with peritoneal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
MRSA bacteremia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anaphylaxis after insect bites (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Fall with fracture of right shoulder and right wrist pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
C. Diff Colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
1.) No new radiographs were conducted. 2) No assessment of adherence to home exercise. 3) This study was conducted in one geographic region and only included participants with regular internet access, which may limit generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT02312713/Prot_SAP_000.pdf